CLINICAL TRIAL: NCT04035772
Title: Implementation and Evaluation of a Wiki Involving Multiple Stakeholders Including Patients in the Promotion of Best Practices in Trauma Care: the WikiTrauma Interrupted Time Series Protocol
Brief Title: The WikiTrauma Interrupted Time Series Protocol
Acronym: WikiTrauma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility (barriers to implantation within the institution)
Sponsor: Laval University (Other)
Collaborators: Canadian Medical Protective Association (Other)
Responsible Party: Principal Investigator, Patrick Archambault, Associate Professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Wiki Implementation 1415-041
Record Dates: First submitted 2018-01-18; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Trauma
Keywords: interrupted time series; wiki; quality improvement; knowledge translation; trauma care; stakeholder engagement; adaptating knowledge tools
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wiki101 and WikiTrauma (Experimental): Wiki101, a theory-based continuing professional development (CPD) program, will train participants at the selected trauma centers to use WikiTrauma effectively and safely to create and share different types of Knowledge Transfer (KT) tools (e.g., care protocols, order sets, patient decision aids). Participants will receive Wiki101 training and then gain access to WikiTrauma with editing rights to the knowledge implementation tools (e.g. care protocols, order sets, care pathways) found in the wiki.
  WikiTrauma is the wiki we created to promote best practices in trauma care and will be implemented in four trauma centers in Quebec during 12 months. During this period, we will continue to measure the impact on the quality of care.
  Interventions: Other: Wiki101 and WikiTrauma

INTERVENTIONS:
Other: Wiki101 and WikiTrauma — Wiki101 is a theory-based continuing professional development course to teach healthcare professionals how to use WikiTrauma. WikiTrauma is a wiki containing implementation tools built upon the Google Sites platform.

SUMMARY:
The purpose of this study is to study the combined effect of WikiTrauma, a free collaborative database of clinical decision support tools, and Wiki101, a training course teaching participants how to use WikiTrauma, on the quality of care in four trauma centers in Quebec.

The hypothesis that the theory-based intervention (Wiki101), in combination with use of WikiTrauma, will result in better adoption of best practices in trauma care, safer care (less complications), improved patient outcomes and less costly care in Canada.

DETAILED DESCRIPTION:
Trauma is the most common cause of mortality among people between the ages of 1 and 45 years, costing Canadians 19.8 billion dollars a year (2004 data), yet half of all patients with major traumatic injuries do not receive evidence-based care, and significant regional variation in the quality of care across Canada exists. Accordingly, the goal of this study is to lead a research project in which stakeholders themselves will adapt evidence-based trauma care knowledge tools to the varied institutional contexts and cultures. This will be done by developing and assessing the combined impact of WikiTrauma, a free collaborative database of clinical decision support tools, and Wiki101, a training course teaching participants how to use WikiTrauma. WikiTrauma has the potential to ensure that all stakeholders (eg, patients, clinicians, and decision makers) can all contribute to, and benefit from, evidence-based clinical knowledge about trauma care that is tailored to the needs and clinical setting.

The main goal will be to study the combined effect of WikiTrauma and Wiki101 on the quality of care in four trauma centers in Quebec.

First, the wiki will be pilot-tested with potential users to create a version ready to test in practice. A rapid, iterative prototyping process with 15 health professionals from nonparticipating centers will allow to identify and resolve usability issues prior to finalizing the definitive version for the interrupted time series. Second, an interrupted time series will be performed to measure the impact of the combined intervention on the quality of care in four trauma centers that will be selected;one level I, one level II, and two level III centers. Participants will be health care professionals working in the selected trauma centers. Also, five patient representatives will be recruited to participate in the creation of knowledge tools destined for the use (eg, handouts). All participants will be invited to complete the Wiki101 training and then use, and contribute to, WikiTrauma for 12 months. The primary outcome will be the change over time of a validated, composite, performance indicator score based on 15 process performance indicators found in the Quebec Trauma Registry.

The project was funded in November 2014 by the Canadian Medical Protective Association. The trial will start in early 2015 and preliminary results should be available in June 2016. Two trauma centers have already agreed to participate and two more will be recruited in the next months.

This study is expected to add important and unique evidence about the effectiveness, safety, and cost savings of using collaborative platforms to adapt knowledge implementation tools across jurisdictions.

ELIGIBILITY:
Inclusion Criteria:

* decision makers (eg, trauma program coordinators) or,
* health care professionals (eg, emergency physicians, critical care physicians, trauma surgeons, nurses, respiratory therapists, physiotherapists, or pharmacists).
* Patient representatives will be selected without any restrictions or limitations with regard to the qualifications.
* Health care professional students and trainees (eg, residents, medical students, and nursing students) will have the same access to WikiTrauma and Wiki101 as fully certified professionals.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Composite performance indicator score (change is assessed) | 30 months prior to implementation and up to 12 months later
  Composite performance indicator score based on 15 process performance indicators found in the Quebec Trauma Registry

SECONDARY OUTCOMES:
Rate of complications (change is assessed) | 30 months prior to implementation and up to 12 months later
  Rate of complication in the trauma center
Mortality rate (change is assessed) | 30 months prior to implementation and up to 12 months later
  Mortality rate in the trauma center
Length of stay (change is assessed) | 30 months prior to implementation and up to 12 months later
  Length of stay in the trauma center
Functional Independence Measure (FIM) (change is assessed) | 30 months prior to implementation and up to 12 months later
  an 18-item of physical, psychological and social function

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Archambault, MD MSc FRCPC, Principal Investigator — CISSS Chaudières-Appalaches (Hôtel-Dieu de Lévis)
Locations (1):
- Pascal Y Smith, Lévis, Quebec, Canada